CLINICAL TRIAL: NCT04726722
Title: Evaluation of an Adaptable and Personcentered Internet-based CBT Program Aimed to Treat Stress, Anxiety and Depressive Symptoms in Patients With Cardiovascular Disease
Brief Title: Evaluation of a Personcentered Internet-based CBT Program for Stress, Anxiety and Depressive Symptoms in Patients With Cardiovascular Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Linkoeping (Other)
Responsible Party: Principal Investigator, Peter Johansson, Professor, Linkoeping University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2020-00935
Record Dates: First submitted 2021-01-22; First posted 2021-01-27 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Cardiovascular Disease; Psychological Distress
Keywords: Cardiovascular disease; Psychological distress; Internet-based cognitive behavioural therapy
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: 2 x 2
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Design of the CBT treatment content (Experimental): Patient determined CBT content (i.e. person-centered) vs. therapist determined I-CBT content
  Interventions: Behavioral: internet-based cognitive behavioral theraphy
- Control of support and feedback (Experimental): Patient-controlled support and feedback (person-centred) vs. therapist -controlled.
  Interventions: Behavioral: internet-based cognitive behavioral theraphy

INTERVENTIONS:
Behavioral: internet-based cognitive behavioral theraphy — When determining the content of the I-CBT program, the participants and therapist will be allowed to choose from a library of treatment modules.
  Therapist controlled support and feedback are given weekly and in a structured manner. Participants will be able to contact the therapist when support and feedback is desired

SUMMARY:
To evaluate a nine-week adaptable and person-centred I-CBT program that can be directed towards stress, anxiety and depressive symptoms in persons with CVD.

DETAILED DESCRIPTION:
All patients diagnosed as CVD (i.e. diagnosis Ischemia (ICD-code I20., I25.), Heart Failure (ICD-code I50., I42.) or Arrhythmia (ICD-code I48, I49, DF016) and who received care in the last 12 months at hospitals in the south-east of Sweden will be contacted by letter with information about the study.

Participants who are interested are invited to visit our website for more information, registration and provision of informed consent. After registration, participants will respond to questions about demographics, medical history, stress, anxiety and depressive symptoms on the website. Inclusion or exclusion will be assessed by a group consisting of a psychologist, cardiology specialist nurse and a psychiatry specialist nurse.

Before final inclusion and randomization eligible participants will be contacted for a telephone interview held by the study nurses.

Included (n=400) participants will, on our website (www.xxxxxx), complete the baseline study questionnaires and then be randomized according to a 2 x2 factorial design.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years and above
* treatment for cardiovascular disease (CVD) according to European Society of Cardiology guidelines
* stable CVD (New York Heart Association class I-III) and not having been hospitalised for CVD in in the last four weeks.
* stress (Perceived Stress Scale (PSS)-10>13 points) and/or
* anxiety (i.e. General Anxiety Disorder Scale (GAD) ≥5 points) and/or
* depressive symptoms (Patient Health Questionnaire-9 28 (PHQ-9) > 5 points)

Exclusion Criteria:

* severe CVD (New York Heart Association classification IV) or another severe chronic life-threatening disease
* severe stress, anxiety or depression assessed as requiring acute treatment
* not being able to dedicate 3-4 hours per week to participate in the program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2023-03-13 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Change in stress from baseline to 9 weeks on the 10 item Perceived Stress Scale | From baseline to 9 weeks at the end of the intervention.
  The 10-item Perceived Stress Scale is a valideted self-report of Stress. The instreument measures the degree to which individuals perceives their life situations as stressful. The 10 items are rated on a 5 point scale and higher scores means more stress
Change in anxiety from baseline to 9 weeks on the 7-item Generalized Anxiety Disorder Scale. | From baseline to 9 weeks at the end of the intervention.
  General Anxiety Disorder scale is validagted self-resport that measure symptoms of general anxiety during the last two weeks. The 7-items range from 0 (not bothered at all) to 3 (nearly every day). A higher score indicate more anxiety and the cut-off 5 suggests at least mild anxiety.
Change in depressive symptoms from baseline to 9 weeks on the 9 item Patient Health Questionnaire. | From baseline to 9 weeks at the end of the intervention.
  The 9-item Patient Health Questionnaire is a validated self-report that measure depressive symtpoms during the last two weeks. Each item is answered on a four graded scale where 0 means that the person not is affected and 3 where the person is affected several Days to almost every day. Higher numbers represents higher levels of depressive symptoms. A cut-off >5 represents at least mild depression.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Johansson, Ph.D, Principal Investigator — Department of Health, Medicine and Caring Sciences, Linkoping University
Locations (1):
- Peter Johansson, Norrköping, Linköpings Universitet, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
Our university works with the question of we can share IPD without violoating GPDR